CLINICAL TRIAL: NCT00905008
Title: Long-Term Safety and Efficacy of Drug Eluting Stents in "Real World" - Results From the FReIburger STent Registry
Brief Title: Long-Term Safety of Drug Eluting Stents in the "Real World" (FReIburger STent Registry)
Acronym: FRIST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. Thorsten Grumann, Department of Cardiology and Angiology, University Freiburg
Other Study IDs: FRIST_GH0102
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Stent Thrombosis
Keywords: drug-eluting stent; bare-metal stent; long-term safety; mortality; stent thrombosis; Angioplasty; Transluminal; Percutaneous Coronary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DES: Patients underwent percutaneous coronary intervention and received at least one drug-eluting stent during their index hospitalisation.
  Interventions: Procedure: transluminal percutaneous coronary intervention; Device: Drug-Eluting and Bare-Metal stents
- BMS: Patients underwent percutaneous coronary intervention and received at least one uncoated stent during their index hospitalisation.
  Interventions: Procedure: transluminal percutaneous coronary intervention; Device: Drug-Eluting and Bare-Metal stents

INTERVENTIONS:
Procedure: transluminal percutaneous coronary intervention — All interventions were done according to current practice guidelines. The operator was responsible for the decision to choose a specific treatment strategy. Angiographic success was defined as residual stenosis <30% by visual analysis in the presence of TIMI 3 flow grade. The patients were prescribed aspirin plus clopidogrel 75 mg per day, after a loading dose of 300 mg or 600 mg, before or during the index coronary intervention. After procedure, all patients were advised to maintain lifelong use of aspirin. The use of clopidogrel (75 mg per day) was always adapted according to guideline recommendations. Heparin was infused throughout the procedure to maintain an activated clotting time of at least 250 sec. The administration of platelet glycoprotein IIb/IIIa receptor blocker was encouraged, unless in existing contraindications.
Device: Drug-Eluting and Bare-Metal stents — Sirolimus-eluting stents (Cypher®), Paclitaxel-eluting stents (Taxus®) Zotarolimus-eluting stents (Endeavor®) and uncoated (bare-metal) stents

SUMMARY:
The FReIburger STent Registry (FRIST) is designed to determine the long term safety and efficacy of Drug Eluting Stents (DES) in a "real-world" patient population requiring stent implantation.

FRIST included patients treated with DES and bare-metal stents (BMS) in the University Hospital of Freiburg, Germany, according to a non-restrictive inclusion criterion, in which virtually all consecutive patient subsets were considered eligible.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing percutaneous coronary intervention

Exclusion Criteria:

* Patient refusal or inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: FRIST (FReIburger STent) is a single-centre, long-term stent registry in a high volume tertiary referral cardiovascular centre. FRIST included patients treated with drug-eluting stents and uncoated stents at the University Hospital of Freiburg, Germany, according to non-restrictive inclusion criterions, in which virtually all consecutive patient subsets were considered eligible.
Sampling Method: Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
All cause mortality (cardiac- and non-cardiac death). | 5 years

SECONDARY OUTCOMES:
The composite of death and MI and stent thrombosis. | 5 years
The occurrence of TVR, stroke, major bleeding, sepsis and tumor were also assessed. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Grumann, MD, Principal Investigator — University of Freiburg

REFERENCES:
- [Derived] Kersting S, Grumann T, Hummel J, Hauschke D, Bode C, Hehrlein C. Impact of chronic kidney disease on long-term clinical outcomes after percutaneous coronary intervention with drug-eluting or bare-metal stents. Crit Pathw Cardiol. 2012 Sep;11(3):152-9. doi: 10.1097/HPC.0b013e31825d267a. PMID 22825536